CLINICAL TRIAL: NCT02554279
Title: A Randomized, Assessor-blind Trial Comparing MENOPUR® (Menotropins for Injection) and Recombinant FSH (Follicle Stimulating Hormone) in a GnRH Antagonist Cycle With Single-Blastocyst Transfer in a High Responder Subject Population
Brief Title: MENOPUR® in a Gonadotropin-Releasing Hormone (GnRH) Antagonist Cycle With Single-Blastocyst Transfer in a High Responder Subject Population
Acronym: MEGASET HR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000205
Record Dates: First submitted 2015-09-09; First posted 2015-09-18 (Estimated); Results first posted 2018-03-02 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2019-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins; follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- menotropin (Experimental): menotropins for injection
  Interventions: Drug: menotropin
- recombinant FSH (Active Comparator)
  Interventions: Drug: recombinant FSH

INTERVENTIONS:
Drug: menotropin
  Other Names: Menopur®
  Arms: menotropin
Drug: recombinant FSH
  Other Names: Gonal-f®
  Arms: recombinant FSH

SUMMARY:
The purpose of this trial is to demonstrate non-inferiority of MENOPUR® versus recombinant Follicle Stimulating Hormone (rFSH) (Gonal-f®) with respect to ongoing pregnancy rate in women undergoing controlled ovarian stimulation (COS) following GnRH treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 21 to 35 years with regular ovulatory menstrual cycles of 21 to 45 days, with a Body Mass Index (BMI) between 18 and 30 kg/m2 who desire pregnancy.
* Subjects must be high responders, defined as subjects who have a serum anti-Müllerian hormone (AMH) ≥5 ng/mL at screening.
* Documented history of infertility (e.g., unable to conceive for at least 12 months or for at least 6 months if receiving donor sperm) with a Day 2 or Day 3 serum FSH level between 1 and 12 IU/L (inclusive), the results of which should be obtained within 6 months prior to randomization.

Exclusion Criteria:

* Known stage III-IV endometriosis (American Society for Reproductive Medicine, 2012).
* History of recurrent miscarriage not followed by a live birth (recurrent is defined as two (2) or more consecutive miscarriages).
* Previous in vitro fertilization (IVF) or assisted reproductive technology (ART) failure due to a poor response to gonadotropins. Poor response is defined as development of ≤2 mature follicles or history of 2 previous failed cycle cancellations prior to oocytes retrieval due to poor response.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 620 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (35):
- United States (35):
  - Bloom Reproductive Institute, Scottsdale, Arizona
  - Fertility Treatment Center, Tempe, Arizona
  - HRC Fertility, Encino, California
  - California Fertility Partners, Los Angeles, California
  - Colorado Center for Reproductive Medicine (CCRM), Lone Tree, Colorado
  - Reproductive Associates of Delaware, Newark, Delaware
  - Women's Medical Research Group, Clearwater, Florida
  - Fertility and IVF Center of Miami, Miami, Florida
  - Center for Reproductive Medicine, Orlando, Florida
  - The Reproductive Medicine Group, Tampa, Florida
  - Georgia Reproductive Specialists, Sandy Springs, Georgia
  - Fertility Institute of Hawaii, Honolulu, Hawaii
  - Idaho Center for Reproductive Medicine, Boise, Idaho
  - Fertility Centers of Illinois, Chicago, Illinois
  - InVia Fertility Specialists, SC, Hoffman Estates, Illinois
  - The Advanced IVF Institute, Naperville, Illinois
  - Shady Grove Fertility Centers, Rockville, Maryland
  - Shady Grove Fertility, Towson, Maryland
  - IVF New England, Lexington, Massachusetts
  - Boston IVF, Waltham, Massachusetts
  - Fertility Center of Las Vegas, Las Vegas, Nevada
  - Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey
  - Reach, Charlotte, North Carolina
  - Carolina Conceptions, Raleigh, North Carolina
  - Abington Hospital, Jefferson Health, Abington, Pennsylvania
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Coastal Fertility Specialists, Mt. Pleasant, South Carolina
  - Center for Assisted Reproduction, Bedford, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Utah Fertility Center, Pleasant Grove, Utah
  - Reproductive Care Center, Sandy City, Utah
  - The Jones Institute for Reproductive Medicine, Norfolk, Virginia
  - Virginia Center for Reproductive Medicine, Reston, Virginia
  - Seattle Reproductive Medicine, Seattle, Washington

REFERENCES:
- [Result] Khair A, Brown T, Markert M, Barsoe CR, Daftary GS, Heiser PW. Highly Purified Human Menopausal Gonadotropin (HP-hMG) Versus Recombinant Follicle-Stimulating Hormone (rFSH) for Controlled Ovarian Stimulation in US Predicted High-Responder Patients: A Cost-Comparison Analysis. Pharmacoecon Open. 2023 Sep;7(5):851-860. doi: 10.1007/s41669-023-00429-8. Epub 2023 Jul 22. PMID 37480456
- [Derived] Robins JC, Khair AF, Widra EA, Alper MM, Nelson WW, Foster ED, Sinha A, Ando M, Heiser PW, Daftary GS. Economic evaluation of highly purified human menotropin or recombinant follicle-stimulating hormone for controlled ovarian stimulation in high-responder patients: analysis of the Menopur in Gonadotropin-releasing Hormone Antagonist Single Embryo Transfer-High Responder (MEGASET-HR) trial. F S Rep. 2020 Nov 10;1(3):257-263. doi: 10.1016/j.xfre.2020.09.010. eCollection 2020 Dec. PMID 34223253
- [Derived] Witz CA, Daftary GS, Doody KJ, Park JK, Seifu Y, Yankov VI, Heiser PW; Menopur in GnRH Antagonist Cycles with Single Embryo Transfer - High Responder (MEGASET-HR) Trial Group. Randomized, assessor-blinded trial comparing highly purified human menotropin and recombinant follicle-stimulating hormone in high responders undergoing intracytoplasmic sperm injection. Fertil Steril. 2020 Aug;114(2):321-330. doi: 10.1016/j.fertnstert.2020.03.029. Epub 2020 May 13. PMID 32416978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 infertility centers in the US between 31 Aug 2014 to 02 Feb 2017.
Groups:
- Menotropin: Menotropins for injection, provided as a vial with powder (75 international units [IU] follicle stimulating hormone [FSH] activity and 75 IU luteinizing hormone [LH] activity) and a vial with diluent.
- Recombinant FSH: Follitropin alpha for injection, a human FSH preparation of recombinant deoxyribonucleic acid (DNA) origin, provided as pen and cartridges filled with either 300 or 450 IU of FSH activity.
Period: Overall Study
Arm/Group | Menotropin | Recombinant FSH
Started | 311 | 309
Treated | 310 | 309
Completed Day 6 of Stimulation | 308 | 309
Received Trigger | 293 | 307
Completed Oocyte Retrieval | 292 | 306
Completed Fresh Blastocyst Transfer | 201 | 191
Completed | 279 | 291
Not Completed | 32 | 18
Not completed — Adverse Event | 2 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Protocol Violation | 2 | 1
Not completed — Other reason | 19 | 6

BASELINE CHARACTERISTICS:
Groups:
- Menotropin: Menotropins for injection, provided as a vial with powder (75 IU FSH activity and 75 IU LH activity) and a vial with diluent.
- Recombinant FSH: Follitropin alpha for injection, human FSH preparation of recombinant DNA origin, provided as pen and cartridges filled with either 300 or 450 IU of FSH activity.
- Total: Total of all reporting groups
Arm/Group | Menotropin | Recombinant FSH | Total
Number analyzed (Participants) | 310 | 309 | 619
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (3.08) | 30.4 (3.02) | 30.2 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310 | 309 | 619
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 18 | 33 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 25 | 43
  White | 270 | 244 | 514
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 310 | 309 | 619

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy Rate
Description: Defined as the percentage of participants with the presence of at least 1 intrauterine pregnancy with a detectable fetal heartbeat at 10-11 weeks of gestation.
Time Frame: 8-9 weeks after blastocyst transfer in the fresh cycle
Population: The modified intent-to-treat (mITT) analysis set comprised all randomized participants who received at least 1 dose of investigational medicinal product.
Measure: Number; unit: percentage of participants
Groups:
- Menotropin: Menotropins for injection, provided as a vial with powder (75 IU activity and 75 IU LH activity) and a vial with diluent.
- Recombinant FSH: Follitropin alpha for injection, a human FSH preparation of recombinant DNA origin, provided as pen and cartridges filled with either 300 or 450 IU of FSH activity.
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 310 | 309
percentage of participants | 35.5 | 30.7
Statistical Analysis 1: Comparison: Menotropin vs Recombinant FSH; Null hypothesis was defined as the difference between ongoing pregnancy rate of participants randomized and treated with menotropin and recombinant FSH, as ≤-12%; Test type: Non-Inferiority — The study had at least 80% power, to demonstrate the non-inferiority of menotropin to recombinant FSH at 1-sided significance level of 0.025 with a -12% non-inferiority margin; Absolute difference = 4.7, 95% CI 2-sided [-2.7 to 12.1]

2. Secondary Outcome: Positive β-human Chorionic Gonadotropin (hCG) Rate
Description: Defined as the percentage of participants with 2 positive β-hCG tests within 2 days in serum.
Time Frame: First test approximately 10-14 days after blastocyst transfer in the fresh cycle, with a second test approximately 2 days later if first test was positive
Population: The mITT analysis set comprised all randomized participants who received at least 1 dose of investigational medicinal product.
Measure: Number; unit: percentage of participants
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 310 | 309
percentage of participants | 40.6 | 39.5
Statistical Analysis 1: Comparison: Menotropin vs Recombinant FSH; Test type: Other; Absolute difference = 1.2, 95% CI 2-sided [-6.6 to 8.9]

3. Secondary Outcome: Clinical Pregnancy Rate
Description: Defined as percentage of participants with transvaginal ultrasound (TVUS) showing at least 1 intrauterine gestational sac with fetal heart beat at 6-7 weeks of gestation.
Time Frame: 4-5 weeks after blastocyst transfer in the fresh cycle
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 310 | 309
percentage of participants | 37.1 | 33.3
Statistical Analysis 1: Comparison: Menotropin vs Recombinant FSH; Test type: Other; Absolute difference = 3.8, 95% CI 2-sided [-3.8 to 11.3]

4. Secondary Outcome: Early Pregnancy Loss
Description: Defined as participants with 2 positive β-hCG tests but no ongoing pregnancy at 10-11 weeks of gestation in the fresh cycle. Percentage of participants with early pregnancy loss is presented.
Time Frame: At 10-11 weeks of gestation in the fresh cycle
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 126 | 122
percentage of participants | 14.3 | 23.8
Statistical Analysis 1: Comparison: Menotropin vs Recombinant FSH; Test type: Other; Absolute difference = -9.5, 95% CI 2-sided [-19.2 to 0.2]

5. Secondary Outcome: Follicular Development as Assessed by TVUS
Description: Defined as average follicle size and average size of 3 largest follicles.
Time Frame: On stimulation Day 6 and last day of stimulation (a maximum of 20 stimulation days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Menotropin, Stimulation Day 6: Menotropins for injection at stimulation Day 6. Menotropins for injection, provided as a vial with powder (75 IU FSH activity and 75 IU LH activity) and a vial with diluent.
- Recombinant FSH, Stimulation Day 6: Recombinant FSH at stimulation Day 6. Follitropin alpha for injection, a human FSH preparation of recombinant DNA origin, provided as pen and cartridges filled with either 300 or 450 IU of FSH activity.
- Menotropin, Last Stimulation Day: Menotropin at last stimulation day. Menotropins for injection, provided as a vial with powder (75 IU FSH activity and 75 IU LH activity) and a vial with diluent.
- Recombinant FSH, Last Stimulation Day: Recombinant FSH at last stimulation day. Follitropin alpha for injection, a human FSH preparation of recombinant DNA origin, provided as pen and cartridges filled with either 300 or 450 IU of FSH activity
Arm/Group | Menotropin, Stimulation Day 6 | Recombinant FSH, Stimulation Day 6 | Menotropin, Last Stimulation Day | Recombinant FSH, Last Stimulation Day
Number analyzed (Participants) | 309 | 309 | 278 | 296
mm
  Average follicle size | 5.95 (1.682) | 7.45 (2.044) | 12.20 (3.328) | 13.28 (2.808)
  Average size of 3 largest follicles | 9.69 (3.562) | 12.17 (2.590) | 21.36 (2.524) | 21.09 (2.685)

6. Secondary Outcome: Follicular Development as Assessed by TVUS
Description: Defined as percentage of participants with follicles having a diameter of ≤9 mm, 10-11 mm, 12-14 mm, 15-16 mm, and ≥17 mm.
Time Frame: On stimulation Day 6 and last day of stimulation (a maximum of 20 stimulation days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Menotropin, Stimulation Day 6 | Recombinant FSH, Stimulation Day 6 | Menotropin, Last Stimulation Day | Recombinant FSH, Last Stimulation Day
Number analyzed (Participants) | 309 | 309 | 278 | 296
percentage of participants
  Follicle size ≤9 mm | 99.0 | 96.4 | 78.4 | 69.9
  Follicle size 10-11 mm | 73.8 | 93.2 | 82.7 | 75.7
  Follicle size 12-14 mm | 50.2 | 76.1 | 93.5 | 96.6
  Follicle size 15-16 mm | 12.6 | 24.9 | 84.9 | 96.3
  Follicle size ≥17 mm | 5.2 | 9.7 | 100 | 100

7. Secondary Outcome: Number of Oocytes Retrieved
Time Frame: At oocyte retrieval visit (approximately 36 hours after hCG administration)
Population: The mITT analysis set comprised all randomized participants who received at least 1 dose of investigational medicinal product. The number of participants analyzed represent the participants with oocytes retrieved.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 292 | 306
oocytes | 15.1 (10.12) | 22.2 (11.54)

8. Secondary Outcome: Number of Metaphase II Oocytes
Time Frame: At oocyte retrieval visit (approximately 36 hours after hCG administration)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: metaphase II oocytes
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 292 | 306
metaphase II oocytes | 10.1 (7.18) | 15.9 (9.01)

9. Secondary Outcome: Fertilization Rate
Description: Defined as 100 times the ratio of number of fertilized 2 pronuclei oocytes to the number of oocytes retrieved, for each participant.
Time Frame: On day 1 post-insemination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of each participant
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 289 | 305
percentage of each participant | 55.09 (21.731) | 59.07 (18.731)

10. Secondary Outcome: Quality of Embryos
Description: Assessed by blastomere uniformity, cell size, the degree of fragmentation, and visual signs of multinucleation.
Time Frame: 3 days after oocyte retrieval
Population: as for outcome 2
Measure: Number; unit: percentage of embryos
Units Other Than Participants: Total number of embryos
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 310 | 309
Number analyzed (Total number of embryos) | 2409 | 4028
percentage of embryos
  Blastomere uniformity-Equally sized blastomeres | 63.1 | 59.0
  Cell size classification-Stage specific | 75.5 | 70.8
  Degree of fragmentation-≤10% | 81.1 | 81.0
  Multinucleation present | 0.7 | 1.1

11. Secondary Outcome: Quality of Embryos
Description: Assessed by cleavage stage.
Time Frame: 3 days after oocyte retrieval
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: blastomeres
Units Other Than Participants: Total number of blastomere
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 310 | 309
Number analyzed (Total number of blastomere) | 2380 | 4001
blastomeres | 7.5 (2.28) | 7.4 (2.32)

12. Secondary Outcome: Quality of Blastocysts
Description: Assessed by blastocyst expansion and hatching status, blastocyst inner cell mass grading, and trophectoderm grading. The scoring was based on the classification system by Gardner and Schoolcraft, with additional categories for inner cell mass (degenerative or no inner cell mass) and trophectoderm (degenerative or very large cell).
Time Frame: 5 days after oocyte retrieval
Population: as for outcome 2
Measure: Number; unit: percentage of embryos
Units Other Than Participants: Embryos reaching blastocyst stage
Arm/Group | Menotropin | Recombinant FSH
Number analyzed (Participants) | 310 | 309
Number analyzed (Embryos reaching blastocyst stage) | 1338 | 2075
percentage of embryos
  Excellent quality | 28.3 | 30.7
  Good quality | 26.5 | 22.5
  Neither | 45.1 | 45.8
  Missing | 0.1 | 1.0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of obtaining informed consent until the last visit (end of trial).
Description: Adverse events with onset after start of the first investigational medicinal product administration were considered treatment-emergent and are presented.
Arm/Group | Menotropin | Recombinant FSH
All-Cause Mortality (participants affected / at risk) | 0/310 | 0/309
Serious Adverse Events (participants affected / at risk) | 8/310 | 11/309
Other Adverse Events (participants affected / at risk) | 179/310 | 218/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menotropin (N=310) | Recombinant FSH (N=309)
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 6 | 10
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menotropin (N=310) | Recombinant FSH (N=309)
Abdominal distension (Gastrointestinal disorders) | 25 | 35
Nausea (Gastrointestinal disorders) | 37 | 40
Abdominal pain (Gastrointestinal disorders) | 21 | 24
Constipation (Gastrointestinal disorders) | 22 | 36
Procedural pain (Injury, poisoning and procedural complications) | 71 | 71
Headache (Nervous system disorders) | 29 | 22
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 30 | 66
Vaginal haemorrhage (Reproductive system and breast disorders) | 21 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol: Clinical Trial Protocol (including amendments 1-4) (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT02554279/Prot_001.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT02554279/SAP_000.pdf